CLINICAL TRIAL: NCT07005375
Title: The Effect of Bathing in the Thermal Mineral Water on the Pain and Performance of Athletes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Polyclinic of the Hospitaller Brothers of St. John of God, Budapest (Other)
Responsible Party: Principal Investigator, Tamas Gati, MD, Polyclinic of the Hospitaller Brothers of St. John of God, Budapest
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Medicinal Water and Rowing; NNGYK/GYSZ/3848-8/2024 (Other: NNGYK/GYSZ/3848-8/2024)
Record Dates: First submitted 2025-04-21; First posted 2025-06-05 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain; Fatigue Recovery; Performance Measures
Keywords: low back pain, fatigue; performance
MeSH Terms: conditions — Low Back Pain; Fatigue | interventions — Water; Water Pollution; Mineral Waters

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, single-blind study.
Who Masked: Participant
Masking Description: Randomized, controlled, single-blind study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Athletes/rowing (Active Comparator): Patients were enrolled if they met the inclusion and exclusion criteria. The classification would be based on a randomization list. Measurements, clinical examinations, and evaluation of pain and functional status-related quality of life will be performed before, immediately after the treatments, and 3 months later. One group will bathe in a pool filled with 36°C thermal mineral water of the Palatinus Spa for 3 weeks, 5 days a week, for a total of 15 sessions, 20 minutes per session. Bathing in the thermal mineral water takes place in the medicinal water pool. The control group does not receive balneotherapy. Both groups can continue their usual training plan. The thermal mineral water-treated group and the control group may not receive systemic or locally administered steroid therapy during the study, and the control group may not receive balneotherapy.
  Interventions: Behavioral: thermal mineral water bath
- Athletes (Active Comparator): One group will bathe in a pool filled with 36°C thermal mineral water of the Palatinus Spa for 3 weeks, 5 days a week, for a total of 15 sessions, 20 minutes per session. Bathing in the thermal mineral water takes place in the medicinal water pool. The control group does not receive balneotherapy. Both groups can continue their usual training plan.
  Rowers coming from the surrounding area, with registration at the Hungarian Rowing Federation
  Interventions: Behavioral: thermal mineral water bath

INTERVENTIONS:
Behavioral: thermal mineral water bath — One group will bathe in a pool filled with 36°C thermal mineral water of the Palatinus Spa for 3 weeks, 5 days a week, for a total of 15 sessions, 20 minutes per session. Bathing in the thermal mineral water takes place in the medicinal water pool. The control group does not receive balneotherapy. Both groups can continue their usual training plan.
  Other Names: water; thermal water; mineral water

SUMMARY:
Effect of bathing in the thermal mineral water well on the performance and potential pain of athletes. Randomized, controlled, single-blind study.

DETAILED DESCRIPTION:
In rowing sports, where the same series of movements are repeated thousands of times, the lower lumbar region is the most stressed part. Because of this, even training on an ergometer can cause numerous lower back problems, even among competitors. In addition, rowers use many muscle groups during their sport, for which the beneficial effect of thermal medicinal waters, affecting the entire musculoskeletal system, can be beneficial, and is used for rehabilitation purposes in several countries.

Studies describe the numerous positive effects of bathing in warm water (37-46°C) in increasing blood flow, regulating blood sugar, and even the positive response of the vascular system.

The Palatinus Spa's water supply is provided by the drilled thermal wells of Margit Island of Budapest.

Regarding its type, the medicinal water is a low salt concentration, calcium-magnesium-hydrogen carbonate, chloride, and sulfate medicinal water, which also has a significant fluoride and metasilicic acid content. The total dissolved mineral content is 1205 mg/liter. In the study, we would conduct the clinical trial necessary for the "Margaret Island mineral water" / 37-38 °C / thermal mineral water of the Margitszigeti É. III well to be declared medicinal water.

Research Question Primary objective: Effect of bathing in the "Margaret Island mineral water" thermal mineral water of the Margaret Island III well on the performance and potential pain of athletes. Randomized, controlled, single-blind study.

Secondary objective: To what extent does thermal water treatment lead to a change in the quality of life of those receiving it compared to their initial condition, and what is the magnitude of this change compared to the control group?

ELIGIBILITY:
Inclusion Criteria:

* Rowers coming from the surrounding area, with registration at the Hungarian Rowing Federation (MESZ), including competitive/touring and recreational/masters rowers
* Women and men between 18 and 75 years of age
* Participating in regular training for at least 6 months
* Signed informed consent form prior to the start of the study

Exclusion Criteria:

* Acute pain;
* Organic neurological deficit;
* Malignancy in the background;
* Pain attributable to inflammatory disease;
* Participants must not have received systemic or local steroid therapy, physiotherapy as a course of treatment, massage therapy, or balneotherapy as a course of treatment within 3 months prior to the study;

General contraindications of balneotherapy:

* unstable angina pectoris,
* uncontrolled hypertension,
* cardiac decompensation,
* respiratory failure,
* unbalanced endocrinological disease,
* acute febrile condition,
* infectious skin diseases,
* other serious internal, urogenital, and other diseases, urinary and fecal incontinence,
* decompensated psychosis and neurosis, lack of compliance

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The extent of the effect and change on the performance of athletes and any existing pain in the balneotherapy group compared to the change in the control group. This would be measured by the improvement in 6000-meter ergometer performance. | 3 months
  The extent of the effect and change on the performance of athletes and any existing pain in the balneotherapy group compared to the change in the control group. This would be measured by the improvement in 6000-meter ergometer performance. Examining the change in threshold load with improving parameters and heart rate variability (HRV) (examining how the heart is able to continuously change the duration between heartbeats (RR intervals) in response to changes in internal and external environmental loads, and thereby showing the heart's adaptation. This adaptability of the heart is based on the optimal interplay and cooperation of the sympathetic and parasympathetic nervous systems.)

SECONDARY OUTCOMES:
The extent of the change in fatigue, muscle pain, and discomfort between workouts measured by VAS in the balneotherapy group compared to the change in the control group. | 3 months
  The extent of the change in fatigue, muscle pain, and discomfort between workouts measured by 1-10 points on a VAS in the balneotherapy group compared to the change in the control group. Change in lumbar spine movement function in cm. Specific questionnaire for lower back pain (Oswestry) Quality of life questionnaire (EuroQuol-5D-5L) Change in medication therapy used for pain. The extent of change on the Borg scale 0-10 points (How much did you exert yourself?)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Budai Irgalmasrendi Kórház Nonprofit Kft., Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No